CLINICAL TRIAL: NCT03631888
Title: Ultrasound Visceral Slide Test for Prediction of Periumblical Adhesions Before Gynecologic Laparoscopic Surgery: a Prospective Cohort Study
Brief Title: Ultrasound Visceral Slide Test for Prediction of Periumblical Adhesions Before Gynecologic Laparoscopic Surgery
Status: Completed | Type: Observational
Sponsor: Barzilai Medical Center (Other)
Responsible Party: Principal Investigator, Ahmad Namazov, Principal investigator, Barzilai Medical Center
Other Study IDs: BRZ 0024-18 CTIL
Record Dates: First submitted 2018-08-12; First posted 2018-08-15 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Periumbilical Adhesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients scheduled for elective laparoscopic surgery
  Interventions: Diagnostic Test: preoperative abdominal ultrasound examination

INTERVENTIONS:
Diagnostic Test: preoperative abdominal ultrasound examination — Performing preoperative abdominal ultrasound examination in patients that will be scheduled for elective laparoscopic surgery for any gynecologic indication

SUMMARY:
Ultrasound visceral slide test for prediction of periumbilical adhesions before gynecologic laparoscopic surgery: a prospective cohort study.

The investigators are planning to conduct a prospective study to evaluate if there is an effect of abdominal wall thickness and body mass index on slide distance of visceral organ during ultrasound examination.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective laparoscopic surgery for any gynecologic indication.

Exclusion Criteria:

* Emergency laparoscopic surgery
* Patients under age 18

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled for elective laparoscopic surgery for any gynecologic indication.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2020-07-12 (Actual); Study Completion 2020-07-27 (Actual)

PRIMARY OUTCOMES:
Visceral Slide Test | 2 minutes
  correlation between abdominal wall thickness(mm) and sliding distance of visceral organ(mm) during ultrasound examination

CONTACTS AND LOCATIONS:
Locations (1):
- Barzilai University Medical Center, Ashkelon, Israel

REFERENCES:
- [Background] Champault G, Cazacu F, Taffinder N. Serious trocar accidents in laparoscopic surgery: a French survey of 103,852 operations. Surg Laparosc Endosc. 1996 Oct;6(5):367-70. PMID 8890421
- [Background] Chapron CM, Pierre F, Lacroix S, Querleu D, Lansac J, Dubuisson JB. Major vascular injuries during gynecologic laparoscopy. J Am Coll Surg. 1997 Nov;185(5):461-5. PMID 9358090
- [Background] Fuller J, Ashar BS, Carey-Corrado J. Trocar-associated injuries and fatalities: an analysis of 1399 reports to the FDA. J Minim Invasive Gynecol. 2005 Jul-Aug;12(4):302-7. doi: 10.1016/j.jmig.2005.05.008. PMID 16036187
- [Background] Brill AI, Nezhat F, Nezhat CH, Nezhat C. The incidence of adhesions after prior laparotomy: a laparoscopic appraisal. Obstet Gynecol. 1995 Feb;85(2):269-72. doi: 10.1016/0029-7844(94)00352-E. PMID 7824244
- [Background] Levrant SG, Bieber EJ, Barnes RB. Anterior abdominal wall adhesions after laparotomy or laparoscopy. J Am Assoc Gynecol Laparosc. 1997 May;4(3):353-6. doi: 10.1016/s1074-3804(05)80227-0. PMID 9154785
- [Background] Ahmad G, O'Flynn H, Duffy JM, Phillips K, Watson A. Laparoscopic entry techniques. Cochrane Database Syst Rev. 2012 Feb 15;(2):CD006583. doi: 10.1002/14651858.CD006583.pub3. PMID 22336819
- [Background] Kodama I, Loiacono LA, Sigel B, Machi J, Golub RM, Parsons RE, Justin J, Zaren HA, Sachdeva AK. Ultrasonic detection of viscera slide as an indicator of abdominal wall adhesions. J Clin Ultrasound. 1992 Jul-Aug;20(6):375-80. doi: 10.1002/jcu.1870200603. PMID 1328308
- [Background] Tu FF, Lamvu GM, Hartmann KE, Steege JF. Preoperative ultrasound to predict infraumbilical adhesions: a study of diagnostic accuracy. Am J Obstet Gynecol. 2005 Jan;192(1):74-9. doi: 10.1016/j.ajog.2004.07.034. PMID 15672006
- [Background] Larciprete G, Valli E, Meloni P, Malandrenis I, Romanini ME, Jarvis S, Rossi F, Barbati G, Cirese E. Ultrasound detection of the "sliding viscera" sign promotes safer laparoscopy. J Minim Invasive Gynecol. 2009 Jul-Aug;16(4):445-9. doi: 10.1016/j.jmig.2009.03.023. PMID 19573821
- [Background] Nezhat CH, Dun EC, Katz A, Wieser FA. Office visceral slide test compared with two perioperative tests for predicting periumbilical adhesions. Obstet Gynecol. 2014 May;123(5):1049-1056. doi: 10.1097/AOG.0000000000000239. PMID 24785858
- [Background] Wilson A, Longhi J, Goldman C, McNatt S. Intra-abdominal pressure and the morbidly obese patients: the effect of body mass index. J Trauma. 2010 Jul;69(1):78-83. doi: 10.1097/TA.0b013e3181e05a79. PMID 20622581
- [Background] Pelosi P, Quintel M, Malbrain ML. Effect of intra-abdominal pressure on respiratory mechanics. Acta Clin Belg. 2007;62 Suppl 1:78-88. PMID 17469705